CLINICAL TRIAL: NCT00877305
Title: Effect of Remote Ischemic Preconditioning on Cognitive Function After Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Patrick Meybohm (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor-Investigator, Patrick Meybohm, PD Dr., University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A165/08
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Cardiac Surgery
Keywords: Ischemic Preconditioning; Cognitive function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC (Active Comparator): Remote Ischemic Preconditioning
  Interventions: Procedure: Remote Ischemic Preconditioning
- CONTROL (Placebo Comparator): Control
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — RIPC will be induced during anesthesia by four 5-min cycles of upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to 200 mmHg (at least a pressure 15 mm Hg greater than the systolic arterial pressure measured via the arterial line).
  Arms: RIPC
Other: Control — Sham intervention with four 5-min cycles of inflation of the blood pressure cuff at 20 mmHg and 5 min deflation without any upper leg ischaemia.
  Arms: CONTROL

SUMMARY:
The purpose of this study is to evaluate the effects of Remote Ischemic Preconditioning on cognitive function in patients undergoing cardiac surgery compared to control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing heart surgery on cardiopulmonary bypass

Exclusion Criteria:

* Emergency cases
* Myocardial infarction up to 7 days prior to enrollment
* Stroke up to 2 months prior to enrollment
* Ejection fraction less than 30%
* Previous psychiatric and neurological illness
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is postoperative neurocognitive dysfunction. | Preoperative, 1 week and 3 months after surgery

SECONDARY OUTCOMES:
New onset of atrial fibrillation, myocardial and kidney injury, cardiac function (previous NCT00882622 study). | Within 24-48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, MD, Principal Investigator — University Hospital Schleswig-Holstein; Berthold Bein, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Kiel, Germany

REFERENCES:
- [Derived] Zitta K, Meybohm P, Bein B, Gruenewald M, Lauer F, Steinfath M, Cremer J, Zacharowski K, Albrecht M. Activities of cardiac tissue matrix metalloproteinases 2 and 9 are reduced by remote ischemic preconditioning in cardiosurgical patients with cardiopulmonary bypass. J Transl Med. 2014 Apr 8;12:94. doi: 10.1186/1479-5876-12-94. PMID 24712447
- [Derived] Meybohm P, Renner J, Broch O, Caliebe D, Albrecht M, Cremer J, Haake N, Scholz J, Zacharowski K, Bein B. Postoperative neurocognitive dysfunction in patients undergoing cardiac surgery after remote ischemic preconditioning: a double-blind randomized controlled pilot study. PLoS One. 2013 May 31;8(5):e64743. doi: 10.1371/journal.pone.0064743. Print 2013. PMID 23741380